CLINICAL TRIAL: NCT00601003
Title: A Phase II Trial of Nifurtimox for Refractory or Relapsed Neuroblastoma or Medulloblastoma.
Brief Title: Study of Nifurtimox to Treat Refractory or Relapsed Neuroblastoma or Medulloblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V0706
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma; Medulloblastoma
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma | interventions — Nifurtimox; Cyclophosphamide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nifurtimox (Experimental)
  Interventions: Drug: Nifurtimox; Drug: Cyclophosphamide; Drug: Topotecan

INTERVENTIONS:
Drug: Nifurtimox — 30mg/kg/day PO divided into TID dosing q day
  Other Names: Lampit
Drug: Cyclophosphamide — 250 mg/m2/dose in normal saline, IV, infused over 30 minutes on days 1-5 of each cycle.
  Other Names: Cytoxan
Drug: Topotecan — 0.75mg/m2/dose, in normal saline, IV, infused over 30 minutes on days 1-5 of each cycle.
  Other Names: Hycamptin

SUMMARY:
The purpose of this study is to determine whether nifurtimox in combination with cyclophosphamide and topotecan are effective in the treatment of relapsed or refractory neuroblastoma and medulloblastoma.

DETAILED DESCRIPTION:
This study is being done to test the effect of a drug, nifurtimox, against neuroblastoma and medulloblastoma in children. Nifurtimox is a drug that has been used in South America for many years to treat a parasitic disease known as Chagas Disease. It is not approved by the Food and Drug Administration for routine use in neuroblastoma or medulloblastoma in the United States, but limited early observations suggest that nifurtimox may have anti tumor activity for neuroblastoma and medulloblastoma.

From the preliminary trials of nifurtimox we have determined a safely tolerated dose of nifurtimox to use in neuroblastoma patients (30mg/kg/day). The dose determined in the Phase I study to be safe, will be the dose used for this study. From clinical experience in South America, we know that children can tolerate nifurtimox when given by mouth, and it appears to have no long-term side effects when used to treat Chagas Disease. Based on our laboratory and animal studies, we believe that drug levels similar to those used to treat Chagas Disease may shrink/kill neuroblastoma cells, especially when combined with other chemotherapy drugs. We do not know whether nifurtimox will shrink/kill tumor cells effectively in children. Therefore, the major goal of the study is to learn if nifurtimox in combination with other chemotherapy drugs is effective in shrinking/killing neuroblastoma and medulloblastoma cells.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-21 years at the time of diagnosis.
* Diagnosis: Histologic verification at either the time of original diagnosis or relapse of neuroblastoma or medulloblastoma.
* Disease Status: Refractory or first or multiple relapsed neuroblastoma, or medulloblastoma that has relapsed after, or is refractory to, a chemotherapy-containing treatment regimen.
* Measurable disease, including at least one of the following:

  * Measurable tumor by CT or MRI
  * For neuroblastoma patients only, a positive MIBG (MIBG not required if subject's neuroblastoma is previously determined to not uptake MIBG), abnormal urinary catecholamine levels, or positive bone marrow biopsy/aspirate.
  * For medulloblastoma patients only, positive CSF cytology
* Current disease state must be one for which there is currently no known curative therapy.
* A negative urine pregnancy test is required for female participants of child bearing potential (≥13 years of age).
* Organ Function Requirements Patients without bone marrow metastases must have an ANC > 500/μl and platelet count >50,000/μl.
* Patients must have adequate liver function as defined by AST or ALT <10x normal
* Informed Consent: All patients and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Life expectancy <2 months or Lansky score <50%
* Investigational Drugs: Patients who are currently receiving another investigational drug are excluded from participation.
* Anti-cancer Agents: Patients who are currently receiving other anticancer agents are not eligible. Patients must have fully recovered from the effects of prior chemotherapy, generally at least 3 weeks from the most recent administration (6 weeks for nitrosoureas).
* Infection: Patients who have an uncontrolled infection are not eligible until the infection is judged to be well controlled.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Compensation for travel related expenses may be available

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2008-01-14 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (15):
- United States (15):
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tufts Medical Center, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics on Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Medical Center, Dallas, Texas
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — http://www.beatcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nifurtimox
Started | 112
Completed | 76
Not Completed | 36

BASELINE CHARACTERISTICS:
Population: Number of subjects that signed consent and had baseline information collected
Arm/Group | Nifurtimox
Number analyzed (Participants) | 112
Age, Continuous [Mean (Full Range); unit: years] | 5.5 [1.1 to 21.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 11
  White | 89
  More than one race | 2
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Related Adverse Events as a Measure of Safety and Tolerability
Description: Test the safety of nifurtimox in children with relapsed or refractory neuroblastoma or medulloblastoma in combination with cyclophosphamide/topotecan
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox
Number analyzed (Participants) | 110
Participants | 45

2. Primary Outcome: Best Radiological Response in Participants Using the RECIST Criteria
Description: Test the efficacy of nifurtimox in children with relapsed or refractory neuroblastoma or medulloblastoma in combination with cyclophosphamide/topotecan
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions, Overall Best Response assessed by CT or MRI, MIBG, and Bone Marrow: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, bone marrow with CR, and MIBG with CR/PR. Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nifurtimox
Number analyzed (Participants) | 76
Participants
  Complete Response | 7
  Partial Response | 11
  Stable Disease | 35
  Progressive Disease | 23

ADVERSE EVENTS:
Time Frame: From first dose of Nifurtimox through to 30 days after last dose, an average of 8 months. Additionally all events deemed related to Nifurtimox were followed past the 30 days to resolution or baseline.
Arm/Group | Nifurtimox
All-Cause Mortality (participants affected / at risk) | 19/110
Serious Adverse Events (participants affected / at risk) | 25/110
Other Adverse Events (participants affected / at risk) | 45/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nifurtimox (N=110)
Anorexia (Gastrointestinal disorders) | 1
Other (Progressive Disease) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17
Sepsis (Infections and infestations) | 2
Nausea and vomiting (Gastrointestinal disorders) | 1
Bladder Thrombosis (Renal and urinary disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Tooth Pain (General disorders) | 1
Seizure (Nervous system disorders) | 3
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Appendicitis (Surgical and medical procedures) | 1
Brain hemorrhage (Vascular disorders) | 1
Aphasia (Nervous system disorders) | 1
Gait Disturbance and Confusion (Nervous system disorders) | 1
confusion/psychosis and dysphagia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nifurtimox (N=110)
Anemia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Ataxia (Nervous system disorders) | 10
Confusion (Nervous system disorders) | 6
Memory Impairment (Nervous system disorders) | 3
Motor Neuropathy/Weakness (Nervous system disorders) | 7
Peripheral Sensory Neuropathy (Nervous system disorders) | 4
Seizures (Nervous system disorders) | 5
ALT elevation (Investigations) | 3
Anorexia (Gastrointestinal disorders) | 7
Febrile Neutropenia (Blood and lymphatic system disorders) | 5
Nausea (Gastrointestinal disorders) | 6
Pain (General disorders) | 4
Vomiting (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT00601003/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT00601003/ICF_001.pdf